CLINICAL TRIAL: NCT00860379
Title: The Effect of Selenium Supplementation Among Pediatric Patients With Burns
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to a shift in primary responsibilities, the PI was not longer able to enroll subjects.
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Maggie Dylewski, PhD,RD, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2007-P-001176
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Results first posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Selenium1 (Experimental): Subject will receive 2 ug/kg of IV selenium per day
  Interventions: Drug: Selenium1
- Selenium2 (Experimental): Subject will receive 4 ug/kg of IV selenium per day
  Interventions: Drug: Selenium2

INTERVENTIONS:
Drug: Selenium1 — 2 ug/kg
  Arms: Selenium1
Drug: Selenium2 — 4 ug/kg
  Arms: Selenium2
Drug: Placebo — IV saline as placebo
  Other Names: saline
  Arms: Placebo

SUMMARY:
The selenium status of children with major burns is suboptimal which may increase the incidence of infection. Se requirements during critical illness are not known. Results from this investigation may provide a tool for recommending Se supplements during burn injury.

The hypothesis of this research is that Se supplementation will restore the depressed Se status among children with burn injuries. The secondary hypothesis is that Se status is related to the incidence of infection among pediatric patients with burns.

DETAILED DESCRIPTION:
Study Title: The effect of selenium supplementation among pediatric patients with burns

Primary Investigator: Maggie L. Dylewski, PhD, RD

Co-investigators: RL. Sheridan, MD; C Ryan, MD; K Prelack, PhD,RD; M Lydon, RN; J Weber, RN, BSN, CIC

Approved by: FDA (IND # 78963), Partners IRB (#2007-P-001176).

Funding: private grant from the Boston Burn Foundation

Background Information: Selenium, an essential dietary nutrient, is a component of glutathione peroxidase (an antioxidant) and thioredoxin reductase, an enzyme that regulates cytokine expression and thus plays a role in the immune system. Previous studies among adult burn patients showed that IV selenium supplementation was related to decreased infection and mortality. Please refer to the study protocol for further details.

Previous Research: We previously showed that children with burns (n = 20) > 20% TBSA had low plasma selenium values compared to reference data of healthy American children. Results from this study also found a significant relationship between plasma selenium and incidence of infections.

Study Design: Randomized, double-blind, placebo-controlled clinical trial

Specific Aims:

1. to determine the impact of supplemental selenium on plasma selenium, glutathione peroxidase activity, and urine selenium among pediatric patients with burns >20% total body surface area (TBSA) burn.
2. to determine the association between selenium supplementation, biomarkers of Se status and indicators of stress and infection.

Subjects: N = 75 pediatric patients with burns.

Inclusion criteria:

* Between 1 and 18 years of age admitted to Shriners Burns Hospital
* TBSA burn of > 20%
* Existing IV catheter
* Enrolled into study within 3 weeks of burn injury

Treatment:

All subjects will be randomized into 1 of 3 groups and receive the treatment for 8 weeks, until 95% wound closure, or until central venous catheter access is discontinued.

1. Placebo (IV 0.9% sodium chloride)
2. 2 mcg/kg/day IV Selenium
3. 4 mcg/kg/day IV Selenium

Biological sample collection:

* 4 mL or 8 mL (8 every other week) of plasma once a week
* 24-hour urine collection once a week

Sample analyses:

* Samples will be frozen until analyses
* Samples will be sent to the outside lab for analyses.
* Plasma will also be sent to Massachusetts General Hospital every other week for plasma selenium analysis (to assess for toxicity)

Primary outcome measures:

* Plasma selenium
* Plasma glutathione peroxidase
* Urine selenium

Secondary outcome measures:

• occurrence of pneumonia or infection (bacterial or fungal) in the wound, blood, or urine

Risks:

* Supplement doses were determined using data from previous studies, current recommended dietary allowance (RDA) and upper tolerable limits, American Society for Parenteral and Enteral Nutrition (ASPEN) guidelines for parenteral selenium, and dietary data recorded from our previous study. According to reference weights (NHANES III) supplement doses do not exceed the upper tolerable limits for children.
* Selenium toxicity is rare. However plasma will be assessed every other week for selenium levels.

Monitoring and Quality Assurance:

* All subjects will be monitored for any treatment-related adverse events for 2 weeks following discontinuation of the study therapy
* Any adverse events will be reported to the Partners Human Research Committee and the FDA per the guidelines.

An independent Data Safety Monitoring Board, consisting of 4 knowledgeable staff members, will meet 2 times per year to monitor the data for safety.

ELIGIBILITY:
Inclusion Criteria:

* Between 1 and 18 years of age admitted to Shriners Burns Hospital
* TBSA burn of > 20%
* Existing IV catheter
* Enrolled into study within 3 weeks of burn injury

Exclusion Criteria:

* < 1 year or > 18 years of age
* < 20% TBSA burn
* No existing IV catheter
* Pre-existing or acute renal disease (creatine > 1.5 mg/dl)
* Pre-existing or acute liver disease (bilirubin > 3)
* Pre-existing or acute thyroid disorders
* Cancer
* AIDS
* Pregnancy (as determined by routine admission labs)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2009-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maggie L Dylewski, PhD,RD, Principal Investigator — Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Selenium 2 ug/kg: Subject will receive 2 ug/kg of IV selenium per day
  Selenium1: 2 ug/kg
- Selenium 4 ug/kg: Subject will receive 4 ug/kg of IV selenium per day
  Selenium2: 4 ug/kg
Period: Overall Study
Arm/Group | Placebo | Selenium 2 ug/kg | Selenium 4 ug/kg
Started | 4 | 6 | 4
Completed | 4 | 6 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Selenium1 | Selenium2 | Total
Number analyzed (Participants) | 4 | 6 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.8 (0.66) | 4.3 (4.0) | 6.3 (5.39) | 4.74 (3.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7
  Male | 2 | 3 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 4 | 6 | 2 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 4 | 14
Total Body Surface Area (TBSA) burn injury [Mean (Standard Deviation); unit: % of body surface area burn] | 48.5 (9.29) | 42.8 (23.16) | 49.3 (26.25) | 46.25 (19.88)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Selenium
Description: plasma selenium of all subjects was assessed
Time Frame: Average plasma selenium calculated over 8 weeks, assessed weekly.
Population: pediatric burn patients
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Selenium1 | Selenium2
Number analyzed (Participants) | 4 | 6 | 4
ng/mL | 45 (5.2) | 46 (19.1) | 52.9 (12.6)

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events between baseline and 2 weeks following discontinuation of the study therapy, up to 10 weeks
Arm/Group | Placebo | Selenium1 | Selenium2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT00860379/Prot_SAP_000.pdf